CLINICAL TRIAL: NCT03566771
Title: Treatment Results and Health Care Consumption From a Web-based CLinical Obesity Support System (CLOSS) - A Randomized Multicentre Trial of Childhood Obesity Treatment
Brief Title: Treatment Results and Health Care Consumption From a Web-based Support System in Behavioural Childhood Obesity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOSS200
Record Dates: First submitted 2018-06-07; First posted 2018-06-25 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Childhood Obesity
Keywords: Mobile Health; Self-Monitoring; Behavioural Treatment
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care according to regular treatment routines at the clinic during 12 months
  Interventions: Behavioral: Usual care
- CLOSS (Active Comparator): Usual care plus using a web-based support system for self-monitoring weight, physical activity and communication with the clinic during 12 months
  Interventions: Behavioral: CLOSS

INTERVENTIONS:
Behavioral: Usual care — The child and parent(s) at regular visits to the pediatric clinic for childhood obesity treatment
  Arms: Usual care
Behavioral: CLOSS — Usual care plus using mobile applications to register weight and physical activity as well as for communication with the clinic. A web-based support system enables health care professionals to follow the patient's daily objectively measured weight and physical activity online.
  Arms: CLOSS

SUMMARY:
This study aims to evaluate if a web-based support system with daily self-monitoring of weight, use of an activity measuring wrist-band, and communication between the clinic and the parents gives better results on degree of obesity compared with usual care. Changes in BMI standard deviation score (SDS) are compared between usual care (control) and usual care with complementary web-based support system (intervention).

DETAILED DESCRIPTION:
In this study children with obesity will be randomized to either usual care according to regular routine (control) or to usual care plus a web-based support system (intervention). Based on previous reviews on mobile health and obesity in combination with the investigators' experiences of childhood obesity treatment components were identified which the researchers hypothesize are of major importance for a web-based system for childhood obesity treatment: Frequent self-monitoring of weight and physical activity, goals for weight loss, and feedback from the treatment team. The system is based on a smart phone application connected to a scale and an activity measuring wrist-band. Data is automatically transferred from the accessories to the smart phone, where data is presented graphically. The data is further transferred to the clinic for support and communication between the clinic and the parents. The randomization will be done at the start of individual treatment and will last for 12 months. The main aim is to evaluate if use of the web-based support system will give better results on degree of obesity compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Obesity according to International Obesity Task Force (IOTF)
* Swedish speaking parents
* Parents able to use a smart phone
* Patients new in treatment or in treatment during the past 9-15 months with a decrease of BMI SDS with ≤0.25

Exclusion Criteria:

* Diagnosed with or undergoing assessment of neuropsychiatric disorder
* Hypothalamic obesity
* Pharmacological treatment that could intervene the obesity treatment

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Changes in degree of obesity | 6 and 12 months after baseline
  Measured by BMI standard deviation score control vs intervention

SECONDARY OUTCOMES:
Number of physical visits | During the intervention 12 months
  Control vs intervention
Cancelation of physical visits | During the intervention 12 months
  Control vs intervention
Time consumption for the health care professionals | During the intervention 12 months
  Time for physical visits, communication and documentation reported by health care professionals. Control vs intervention
Parental experience of treatment | During the intervention 3, 6 and 12 months
  Measured by web-based CLOSS specific questions. Control vs intervention
Health care professional's experiences using the web-based support system | During the intervention 3, 6 and 12 months
  CLOSS specific questions regarding the application
Physical activity level | During the intervention 12 months
  Measured by time and intensity through the activity measuring wrist-band. Only intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson, PhD, Principal Investigator — Karolinska Institutet
Locations (10):
- Sweden (10):
  - Outpatient pediatric clinic at Hisingen, Gothenburg
  - Outpatient pediatric clinic in Kungshöjd, Gothenburg
  - Outpatient pediatric clinic at Hässleholm hospital, Hässleholm
  - Outpatient pediatric clinic at Helsingborg hospital, Helsingborg
  - Outpatient pediatric clinic, Hälsan Barnmottagning, Jönköping
  - Outpatient pediatric clinic at Karlstad hospital, Karlstad
  - Outpatient pediatric clinic at Nacka hospital, Stockholm
  - Pediatric clinic, Umeå University Hospital, Umeå
  - Outpatient pediatric clinic at Västerås central hospital, Västerås
  - Outpatient pediatric clinic at Ystad hospital, Ystad